CLINICAL TRIAL: NCT01813721
Title: Study to Investigate Which Clinical Risk Factors Are Considered by Physicians When Conducting Overall Febrile Neutropenia Risk Assessments for Patients Receiving Chemotherapy With an Intermediate (10% - 20%) Febrile Neutropenia Risk.
Brief Title: Study Investigating How Physicians Assess the Risk of Patients Developing Febrile Neutropenia During Chemotherapy.
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20110146
Record Dates: First submitted 2013-01-08; First posted 2013-03-19 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Chemotherapy-induced Febrile Neutropenia
Keywords: NHL; Breast Cancer; Lung Cancer
MeSH Terms: conditions — Chemotherapy-Induced Febrile Neutropenia; Breast Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: All patients enrolled

SUMMARY:
This is a prospective observational study investigating how physicians assess the risk of febrile neutropenia (FN) developing in patients who will receive chemotherapy.

Approximately 150-200 investigators will take part in about 100 sites in Europe, Canada and Australia. Approximately 1000 subjects will be studied, all of whom will have non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC), non-Hodgkin's lymphoma (NHL) or breast cancer and will be due to receive one of the specific chemotherapy regimens of interest.

Investigators' approach to FN risk assessment will be studied using lists of possible risk factors they may consider during their assessment. Investigators will be asked to select and rank the factors they consider the most important when assessing the overall FN risk of a subject and when making the decision whether to treat with granulocyte-colony stimulating factor (G-CSF) primary prophylaxis (PP). They will be asked to make these selections based initially on their own routine clinical practise and subsequently relating specifically to each subject recruited.

This is a non-interventional study that involves no procedures outside normal care for the subjects; all data collection will be completed prior to chemotherapy administration.

DETAILED DESCRIPTION:
Although a formal hypothesis will not be tested in this observational study, it is hypothesized that the clinical risk factors ranked as the most important when conducting FN risk assessments by investigators are aligned with international guidelines and published data. Also, that the investigator's decision to treat with G-CSF PP is influenced by clinical and non-clinical risk factors (such as distance from site, estimated subject compliance, and access to fully reimbursed G-CSF).

Study Design: Prior to identifying eligible subjects, Investigators will be registered and will record baseline information. During this Baseline Investigator Assessment investigators will be provided with two lists of risk factors. Investigators must rank selected risk factors that they consider to be the most important when assessing 1) overall FN risk (only scientific factors will be included), and 2) when deciding on whether G-CSF PP treatment will be used or not (this list will also contain non clinical factors). They will also record their own FN risk intervention threshold, which is the FN risk threshold score at which they would use G-CSF PP in their usual clinical practice.

Investigators will then prospectively and sequentially identify eligible subjects with NHL, breast or lung cancer who are due to initiate one of the permitted standard dose chemotherapy regimens listed in the protocol. The permitted chemotherapy regimens have an estimated intermediate FN risk (10%-20%) documented in published data and/or international guidelines.

For each enrolled subject, Investigators will complete a Subject Assessment prior to the start of their chemotherapy. They will be provided with the same two lists of risk factors as in the Baseline Assessment and asked to complete them based on each specific subject. Investigators must rank selected risk factors that they consider to be the most important when assessing 1) overall FN risk (only scientific factors will be included), and 2) when deciding on whether G-CSF PP treatment will be used or not. They will also document their final estimated FN risk score as a percentage based on the subject's medical history and standard of care (SOC) assessments (their routine practice for assessing this risk), and a decision as to whether G-CSF PP will be administered. Investigators will record which type of G-CSF they plan to use if one will be used.

End of Study for a subject will occur once these activities have been completed, and a prescription for the first cycle of chemotherapy has been written. The subject data collected will only be historical subject information and laboratory data from SOC assessments performed prior to beginning chemotherapy treatment. No data will be collected after the initiation of chemotherapy.

The approach to the statistical analysis will be generally descriptive in nature. The primary analysis will be conducted at two levels; investigator level and the subject level. It is expected that the opinions of investigators at a single site (that is, a department within a cancer treatment centre) will be correlated. Also, that the opinions about subjects from a single investigator will be more alike than subjects of other investigators; adjustments will be made in the analyses to account for this. Confidence intervals for the investigator level analysis and the subject level data will obtained from Multi-level Modelling (MLM) to allow for the expected intra-site and intra-investigator correlation of investigators within sites and subjects within investigator. In general, categorical data will be summarised by the number and percentage of subjects in each category. Continuous data will be summarised by mean, standard deviation, median, lower and upper quartiles, minimum and maximum values. Two-sided exact 95% confidence intervals (obtained using MLM) will be presented, where appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Any stage NHL, small cell lung cancer (SCLC), non-small cell lung cancer (NSCLC), or breast cancer initiating a new chemotherapy course
* Scheduled to receive one of the permitted standard dose chemotherapy regimens with an estimated intermediate (10%-20%) FN risk according to published data or guidelines (planned dose modifications +/-10% are allowable).
* Before any study-specific procedure, the appropriate written informed consent must be obtained where this is required by local regulations

Exclusion Criteria:

* Ongoing or planned concurrent participation in any clinical study involving Investigational Product that has not been approved by the European Medicines Agency (EMA) or competent authority for any indication,
* Ongoing or planned concurrent participation in any clinical study where the administration of Colony Stimulating Factor (CSF) is determined by the protocol (clinical trials on an approved drug and observational trials are permitted as long as these do not mandate how neutropenia should be treated)
* Prior stem-cell transplantation (includes bone marrow transplantation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects will have NHL, breast or lung cancer and be due to initiate one of the permitted standard dose chemotherapy regimens listed in the protocol (those with a documented intermediate FN risk of 10-20%). Subjects will be prospectively and sequentially identified by approximately 150-200 investigators during their clinics distribututed in 11 countries.
Sampling Method: Probability Sample
Enrollment: 1007 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (79):
- Australia (4):
  - Research Site, Tweed Heads, New South Wales
  - Research Site, Bendigo, Victoria
  - Research Site, Shepparton, Victoria
  - Research Site, Wodonga, Victoria
- Austria (5):
  - Research Site, Eggenburg
  - Research Site, Graz
  - Research Site, Leoben
  - Research Site, Vienna
  - Research Site, Vöcklabruck
- Canada (3):
  - Research Site, Moncton, New Brunswick
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Montreal, Quebec
- France (14):
  - Research Site, Alès Cédex
  - Research Site, Arras
  - Research Site, Besançon
  - Research Site, Brest
  - Research Site, Créteil
  - Research Site, Grenoble
  - Research Site, Marseille
  - Research Site, Montluçon
  - Research Site, Neuilly-sur-Seine
  - Research Site, Nîmes
  - Research Site, Pierre-Bénite
  - Research Site, Saint-Quentin
  - Research Site, Toulon
  - Research Site, Villefranche-sur-Saône
- Germany (8):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Fulda
  - Research Site, Mainz
  - Research Site, Neustadt/Sachsen
  - Research Site, Rostock
  - Research Site, Stralsund
  - Research Site, Twistringen
- Greece (5):
  - Research Site, Athens
  - Research Site, Chania
  - Research Site, Larissa
  - Research Site, Nea Kifissia, Athens
  - Research Site, Thessaloniki
- Ireland (2):
  - Research Site, Cork
  - Research Site, Galway
- Italy (9):
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Foggia
  - Research Site, Monza (MB)
  - Research Site, Pordenone
  - Research Site, Reggio Calabria
  - Research Site, Roma
  - Research Site, Torino
  - Research Site, Varese
- Poland (8):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Elblag
  - Research Site, Gdynia
  - Research Site, Lodz
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (11):
  - Research Site, Brasov
  - Research Site, Brăila
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Focşani
  - Research Site, Iași
  - Research Site, Onești
  - Research Site, Oradea
  - Research Site, Piteşti
  - Research Site, Suceava
  - Research Site, Timișoara
- Spain (10):
  - Research Site, Huelva, Andalusia
  - Research Site, Málaga, Andalusia
  - Research Site, Zaragoza, Aragon
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, San Cristóbal de La Laguna, Canary Islands
  - Research Site, Ávila, Castille and León
  - Research Site, Valladolid, Castille and León
  - Research Site, Barcelona, Catalonia
  - Research Site, Pamplona, Navarre
  - Research Site, Valencia, Valencia

REFERENCES:
- [Background] Freyer G, Kalinka-Warzocha E, Syrigos K, Marinca M, Tonini G, Ng SL, Wong ZW, Salar A, Steger G, Abdelsalam M, DeCosta L, Szabo Z. Attitudes of physicians toward assessing risk and using granulocyte colony-stimulating factor as primary prophylaxis in patients receiving chemotherapy associated with an intermediate risk of febrile neutropenia. Med Oncol. 2015 Oct;32(10):236. doi: 10.1007/s12032-015-0682-z. Epub 2015 Aug 28. PMID 26315712
- [Derived] Lyman GH, Dale DC, Legg JC, Abella E, Morrow PK, Whittaker S, Crawford J. Assessing patients' risk of febrile neutropenia: is there a correlation between physician-assessed risk and model-predicted risk? Cancer Med. 2015 Aug;4(8):1153-60. doi: 10.1002/cam4.454. Epub 2015 Mar 23. PMID 25810005
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on 13 December 2012 and the last patient enrolled on 08 January 2014.
  There were 205 registered investigators, 35 of whom did not enrol any participants and 5 who did not enrol any eligible participants and were excluded from the primary analysis set - investigators (PASI).
Groups:
- All Enrolled Patients: Participants with cancer who were planning to receive standard dose chemotherapy regimens with a documented intermediate risk (10% to 20%) of febrile neutropenia (FN).
Period: Overall Study
Arm/Group | All Enrolled Patients
Started | 1007 (Indicates number of participants enrolled)
Completed | 943
Not Completed | 64
Not completed — Ineligibility determined | 63
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Primary Analysis Set (PAS) is the set of all participants who satisfy the eligibility criteria and had at least one FN risk factor ranked by the investigator in their Subject Assessment.
Arm/Group | Primary Analysis Set
Number analyzed (Participants) | 944
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 554
  Male | 390
Tumor Type [Number; unit: participants]
  Breast cancer | 395
  Non-small cell lung cancer (NSCLC) | 248
  Non-Hodgkin's lymphoma (NHL) | 182
  Small-cell lung cancer (SCLC) | 119
Investigator Specialty [Number; unit: investigators] — Data provided for the Primary analysis Set-Investigators, consisting of the 165 investigators who contributed participants to the primary analysis set.
  investigators
    Medical Oncologist | 110
    Hematologist | 31
    Pulmonologist | 10
    Radiation Oncologist | 8
    Medical Gynecologist | 4
    Gynecological Surgeon | 2
Number of years in oncology/hematology clinical practice [Number; unit: investigators]
  > 10 years | 117
  ≤ 10 years | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Investigators Who Ranked Age and Chemotherapy Regimen as a Risk Factor for Febrile Neutropenia
Description: During the baseline investigator assessment (prior to identification of participants), investigators were provided a list of risk factors on a source document worksheet, and asked to rank the risk factors that they considered to be the most important when assessing overall febrile neutropenia (FN) risk. Age and chemotherapy regimen were specified in the protocol as risk factors of interest. Reported are age and chemotherapeutic agents ranked individually, chemotherapy agents detailed by specific factors, and age and chemotherapy agents jointly ranked. To account for the expected correlation between investigators at the same sites, two-level, empty (no explanatory variables) multilevel models were used in the estimation of the percentages and 95% confidence intervals.
Time Frame: Baseline (prior to participant enrolment)
Population: Primary analysis set - investigators (PASI), which consists of investigators who contributed participants to the primary analysis set (PAS).
Measure: Number (95% Confidence Interval); unit: percentage of investigators
Units Other Than Participants: Investigators
Arm/Group | Primary Analysis Set - Investigators
Number analyzed (Participants) | 944
Number analyzed (Investigators) | 165
percentage of investigators
  Age | 73.4 [64.4 to 80.8]
  Chemotherapy agents in the backbone | 88.3 [81.7 to 92.7]
  Anthracyclines | 41.1 [31.6 to 51.3]
  Taxanes | 25.0 [17.7 to 34.1]
  Platinum(s) | 22.2 [15.1 to 31.6]
  Alkylating agents | 21.5 [14.7 to 30.3]
  Topoisomerase II inhibitors | 13.8 [8.8 to 21.2]
  Topoisomerase I inhibitors | 11.2 [6.8 to 17.8]
  Gemcitabine | 9.7 [5.9 to 15.7]
  Vinorelbine | 9.1 [5.4 to 14.8]
  Other agents | 2.4 [0.9 to 6.4]
  Age and chemotherapy agents in the backbone | 66.3 [57.0 to 74.5]

2. Primary Outcome: Percentage of Investigators Who Ranked Each Factor as a Risk Factor for Febrile Neutropenia (FN)
Description: During the baseline investigator assessment (prior to identification of participants), investigators were provided a list of risk factors on a source document worksheet and asked to rank the risk factors that they considered to be the most important when assessing overall FN risk. To account for the expected correlation between investigators at the same sites, two-level, empty (no explanatory variables) multilevel models were used in the estimation of the percentages and 95% confidence intervals. ECOG = Eastern Cooperative Oncology Group
Time Frame: Assessed at Baseline, prior to participant enrolment.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of investigators
Units Other Than Participants: Investigators
Arm/Group | Primary Analysis Set - Investigators
Number analyzed (Participants) | 944
Number analyzed (Investigators) | 165
percentage of investigators
  Chemotherapy agents in the backbone | 88.3 [81.7 to 92.7]
  History of prior FN | 83.0 [75.7 to 88.5]
  Baseline laboratory values | 76.2 [67.9 to 82.9]
  Age | 73.4 [64.4 to 80.8]
  Prior chemotherapy | 70.5 [62.4 to 77.6]
  Guidelines | 69.9 [60.0 to 78.2]
  Prior radiotherapy involving bone marrow | 64.8 [55.6 to 73.0]
  ECOG/Karnofsky performance status | 64.0 [54.9 to 72.3]
  Tumor type | 62.7 [53.0 to 71.5]
  Comorbidities | 62.5 [53.5 to 70.8]
  Documented bone marrow involvement | 62.4 [51.7 to 72.1]
  Tumor stage | 61.8 [52.8 to 70.2]
  Treatment intent | 50.0 [41.1 to 58.8]
  Nutritional status | 49.2 [40.2 to 58.2]
  Medications taken | 47.9 [38.2 to 57.8]
  Current infection | 45.4 [36.6 to 54.6]
  Concurrent radiotherapy | 42.2 [32.4 to 52.6]
  Personal experience of chemotherapy regimen risk | 40.4 [32.5 to 48.9]
  Open wounds | 37.0 [27.7 to 47.3]
  Planned relative dose intensity | 25.5 [18.2 to 34.6]
  Female gender | 23.2 [15.7 to 32.9]
  Other disease/treatment related | 4.2 [1.9 to 8.9]
  Other patient related | 2.4 [0.9 to 6.4]

3. Primary Outcome: Percentage of Participants for Whom Age and Chemotherapy Regimen Were Ranked as an Important Risk Factor
Description: Investigators ranked the risk factors they considered to be the most important when assessing the overall risk of febrile neutopenia for each participant. Only historical patient information recorded before the beginning of chemotherapy treatment were collected in this study. Age and chemotherapy regimen were specified in the protocol as risk factors of interest. Reported are age and chemotherapeutic agents ranked individually, chemotherapy agents detailed by specific factors, and age and chemotherapy agents jointly ranked. To account for the expected correlation between participants with the same investigators and between investigators at the same sites, three-level, empty (no explanatory variables) multilevel models were used in the estimation of the percentages and 95% confidence intervals.
Time Frame: At enrolment, prior to chemotherapy initiation
Population: Primary analysis set which consists of all participants who satisfied the eligibility criteria and had at least one FN risk factor ranked by the investigator in their Subject Assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Analysis Set
Number analyzed (Participants) | 944
percentage of participants
  Age | 39.4 [31.9 to 47.5]
  Chemotherapy agents in the backbone | 92.6 [88.0 to 95.6]
  Anthracyclines | 36.2 [25.6 to 48.4]
  Taxanes | 17.1 [11.6 to 24.3]
  Platinum(s) | 9.9 [6.4 to 15.1]
  Alkylating agents | 6.9 [4.4 to 10.6]
  Topoisomerase II inhibitors | 2.7 [1.7 to 4.3]
  Vinorelbine | 1.9 [1.1 to 3.4]
  Topoisomerase I inhibitors | 0.1 [0.0 to 0.8]
  Gemcitabine | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model
  Other agents | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model

4. Primary Outcome: Percentage of Participants for Whom Each FN Risk Factor Was Ranked as Important
Description: Investigators ranked the risk factors they considered to be the most important when assessing the overall risk of febrile neutopenia for each participant. Only historical patient information recorded before the beginning of chemotherapy treatment was collected in this study. To account for the expected correlation between participants with the same investigators and between investigators at the same sites, three-level, empty (no explanatory variables) multilevel models were used in the estimation of the percentages and 95% confidence intervals. ECOG = Eastern Cooperative Oncology Group.
Time Frame: At enrolment, prior to chemotherapy initiation.
Population: Primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Analysis Set
Number analyzed (Participants) | 944
percentage of participants
  Chemotherapy agents in the backbone | 92.6 [88.0 to 95.6]
  Tumor type | 72.3 [60.7 to 81.5]
  Guidelines | 61.7 [48.1 to 73.8]
  Tumor stage | 42.9 [33.7 to 52.6]
  Age | 39.4 [31.9 to 47.5]
  Treatment intent | 30.9 [23.7 to 39.1]
  ECOG/Karnofsky performance status | 27.8 [21.2 to 35.5]
  Female gender | 18.4 [12.7 to 25.7]
  Comorbidities | 15.6 [12.3 to 19.7]
  Baseline laboratory values | 15.3 [11.1 to 20.8]
  Personal experience of chemotherapy regimen risk | 15.2 [10.2 to 22.1]
  Prior chemotherapy | 14.8 [11.5 to 18.9]
  Nutritional status | 8.2 [5.8 to 11.5]
  Planned relative dose intensity | 7.1 [4.1 to 11.9]
  Medications taken | 5.2 [3.6 to 7.6]
  History of prior FN | 4.4 [2.9 to 6.5]
  Documented bone marrow involvement | 4.3 [2.7 to 7.0]
  Prior radiotherapy involving bone marrow | 4.0 [2.8 to 5.7]
  Current infection | 3.7 [2.4 to 5.6]
  Concurrent radiotherapy | 2.3 [1.4 to 3.7]
  Open wounds | 2.2 [1.3 to 3.8]
  Other patient related | 2.0 [1.1 to 3.6]
  Other disease/treatment related | 0.8 [0.4 to 1.7]

5. Secondary Outcome: Percentage of Investigators Who Ranked Each Factor in the Granulocyte Colony Stimulating Factor (G-CSF) Primary Prophylaxis (PP) Decision as Important
Description: During the baseline investigator assessment (prior to identification of participants), investigators were provided a list of factors on a source document worksheet, and asked to rank the factors that they considered to be the most important when deciding whether to use G-CSF PP treatment or not. To account for the expected correlation between investigators at the same sites, two-level, empty (no explanatory variables) multilevel models were used in the estimation of the percentages and 95% confidence intervals. ECOG = Eastern Cooperative Oncology Group.
Time Frame: Assessed at baseline, prior to participant enrolment.
Population: Primary analysis set - investigators
Measure: Number (95% Confidence Interval); unit: percentage of investigators
Units Other Than Participants: Investigators
Arm/Group | Primary Analysis Set - Investigators
Number analyzed (Participants) | 944
Number analyzed (Investigators) | 165
percentage of investigators
  Outcome of the overall FN risk assessment | 88.7 [82.6 to 92.9]
  Age | 79.7 [70.6 to 86.5]
  Baseline laboratory values | 73.8 [64.3 to 81.5]
  Guidelines | 70.5 [61.2 to 78.3]
  Treatment intent | 69.4 [60.8 to 76.8]
  ECOG/Karnofsky performance status | 66.1 [56.2 to 74.8]
  Medications taken | 50.8 [40.8 to 60.7]
  Length of chemotherapy cycle | 49.7 [39.0 to 60.3]
  Planned relative dose intensity | 34.2 [25.6 to 44.0]
  Patient lives far from clinic/healthcare resources | 33.8 [25.4 to 43.3]
  Safety risk of intensive chemotherapy | 30.9 [22.7 to 40.4]
  Estimated compliance with the treatment plan | 23.7 [16.8 to 32.3]
  Local access to reimbursed G-CSF PP | 22.7 [15.4 to 32.1]
  Outpatient care of the patient | 20.5 [14.5 to 28.1]
  Safety risk of G-CSFs in general | 19.5 [13.0 to 28.0]
  Hospitalized patient | 16.3 [10.8 to 24.0]
  Family/caregiver/nurse support to the patient | 13.6 [8.3 to 21.3]
  Wait and see approach | 10.2 [6.3 to 16.2]
  Retired vs employed/active status of the patient | 8.5 [4.9 to 14.4]
  Private health insurance of the patient | 6.4 [3.3 to 12.0]
  Other | 0.6 [0.1 to 4.3]

6. Secondary Outcome: Percentage of Investigators Who Ranked Each Factor in the G-CSF PP Decision as Important by Clinical Specialty
Description: During the baseline investigator assessment (prior to identification of participants), investigators were provided a list of factors on a source document worksheet, and asked to rank the factors that they considered to be the most important when deciding whether to use G-CSF PP treatment or not. To account for the expected correlation between investigators at the same sites, two-level, empty (no explanatory variables) multilevel models were used in the estimation of the percentages and 95% confidence intervals. ECOG = Eastern Cooperative Oncology Group. Subgroup analyses were performed where a subgroup contained at least 40 investigators. Results are reported for medical oncologists as this was the only specialty that contained at least 40 investigators.
Time Frame: Assessed at baseline, prior to participant enrolment.
Population: Primary analysis set - investigators; analysis only includes subgroups with at least 40 investigators.
Measure: Number (95% Confidence Interval); unit: percentage of investigators
Units Other Than Participants: Investigators
Arm/Group | Medical Oncologist
Number analyzed (Participants) | 662
Number analyzed (Investigators) | 110
percentage of investigators
  Outcome of the overall FN risk assessment | 88.4 [80.6 to 93.3]
  Treatment intent | 78.5 [69.1 to 85.6]
  Age | 77.7 [66.6 to 86.0]
  Guidelines | 75.5 [65.2 to 83.5]
  Baseline laboratory values | 73.7 [61.5 to 83.1]
  ECOG/Karnofsky performance status | 70.5 [58.2 to 80.4]
  Medications taken | 51.6 [39.2 to 63.9]
  Length of chemotherapy cycle | 46.4 [34.7 to 58.4]
  Planned relative dose intensity | 39.6 [28.8 to 51.6]
  Patient lives far from clinic/healthcare resources | 36.4 [25.7 to 48.7]
  Safety risk of intensive chemotherapy | 28.9 [19.4 to 40.7]
  Estimated compliance with the treatment plan | 27.1 [18.3 to 38.2]
  Local access to reimbursed G-CSF PP | 26.0 [16.4 to 38.7]
  Safety risk of G-CSFs in general | 24.1 [15.2 to 36.0]
  Outpatient care of the patient | 21.9 [14.6 to 31.5]
  Hospitalized patient | 16.4 [9.6 to 26.7]
  Family/caregiver/nurse support to the patient | 13.8 [7.7 to 23.4]
  Retired vs employed/active status of the patient | 10.6 [5.9 to 18.5]
  Wait and see approach | 9.0 [4.8 to 16.4]
  Private health insurance of the patient | 7.1 [3.4 to 14.2]
  Other | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response.

7. Secondary Outcome: Percentage of Investigators Who Ranked Each Factor in the G-CSF PP Decision as Important by Number of Years in Clinical Practice in Oncology / Hematology
Description: During the baseline investigator assessment (prior to identification of participants), investigators were provided a list of factors on a source document worksheet, and asked to rank the factors that they considered to be the most important when deciding whether to use G-CSF PP treatment or not. To account for the expected correlation between investigators at the same sites, two-level, empty (no explanatory variables) multilevel models were used in the estimation of the percentages and 95% confidence intervals. Subgroup analyses were performed where a subgroup contained at least 40 investigators. ECOG = Eastern Cooperative Oncology Group.
Time Frame: Assessed at baseline, prior to participant enrolment.
Population: Primary analysis set - investigators; analysis only includes subgroups with at least 40 investigators.
Measure: Number (95% Confidence Interval); unit: percentage of investigators
Units Other Than Participants: Investigators
Arm/Group | ≤ 10 Years | > 10 Years
Number analyzed (Participants) | 257 | 687
Number analyzed (Investigators) | 48 | 117
percentage of investigators
  Outcome of the overall FN risk assessment | 85.4 [70.6 to 93.4] | 90.2 [82.9 to 94.6]
  Age | 79.2 [61.3 to 90.2] | 79.4 [69.0 to 87.0]
  Guidelines | 77.1 [61.6 to 87.6] | 66.8 [56.0 to 76.1]
  Baseline laboratory values | 69.5 [52.2 to 82.6] | 74.2 [63.6 to 82.6]
  Treatment intent | 64.3 [46.7 to 78.8] | 71.9 [62.0 to 80.0]
  ECOG/Karnofsky performance status | 56.7 [37.9 to 73.7] | 69.7 [58.6 to 79.0]
  Length of chemotherapy cycle | 56.0 [39.2 to 71.6] | 46.7 [34.9 to 58.9]
  Medications taken | 48.2 [31.2 to 65.6] | 51.2 [40.6 to 61.7]
  Safety risk of intensive chemotherapy | 41.2 [24.7 to 60.0] | 27.4 [19.5 to 37.0]
  Patient lives far from clinic/healthcare resources | 39.1 [23.6 to 57.1] | 32.4 [23.7 to 42.5]
  Planned relative dose intensity | 35.5 [21.7 to 52.1] | 33.7 [24.1 to 45.0]
  Local access to reimbursed G-CSF PP | 29.3 [16.9 to 45.8] | 20.7 [12.7 to 32.0]
  Estimated compliance with the treatment plan | 29.1 [17.0 to 45.1] | 22.4 [14.9 to 32.3]
  Safety risk of G-CSFs in general | 24.4 [12.9 to 41.5] | 18.3 [11.5 to 28.0]
  Outpatient care of the patient | 20.8 [10.9 to 36.2] | 20.6 [13.8 to 29.7]
  Family/caregiver/nurse support to the patient | 20.8 [10.9 to 36.2] | 11.5 [6.2 to 20.4]
  Hospitalized patient | 20.7 [10.6 to 36.6] | 15.4 [9.8 to 23.3]
  Retired vs employed/active status of the patient | 14.6 [6.6 to 29.2] | 6.6 [3.1 to 13.2]
  Private health insurance of the patient | 12.5 [5.3 to 26.8] | 4.7 [1.9 to 10.9]
  Wait and see approach | 10.4 [4.0 to 24.4] | 10.3 [5.8 to 17.4]
  Other | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response. | 0.9 [0.1 to 6.1]

8. Secondary Outcome: Percentage of Investigators Who Ranked Each Factor in the G-CSF PP Decision as Important by Institution Type
Description: as for outcome 7
Time Frame: Assessed at baseline, prior to participant enrolment.
Population: Primary analysis set - investigators; analysis only includes subgroups with at least 40 investigators.
Measure: Number (95% Confidence Interval); unit: percentage of investigators
Units Other Than Participants: Investigators
Arm/Group | University Hospital | General Hospital
Number analyzed (Participants) | 302 | 281
Number analyzed (Investigators) | 57 | 46
percentage of investigators
  Outcome of the overall FN risk assessment | 91.9 [79.2 to 97.2] | 84.8 [70.4 to 92.9]
  Baseline laboratory values | 77.5 [56.5 to 90.1] | 71.8 [54.4 to 84.5]
  Age | 75.2 [54.8 to 88.3] | 89.0 [70.9 to 96.4]
  Guidelines | 71.9 [50.2 to 86.7] | 65.1 [46.5 to 80.0]
  Treatment intent | 67.0 [45.6 to 83.1] | 73.9 [58.6 to 85.0]
  ECOG/Karnofsky performance status | 66.3 [50.4 to 79.2] | 71.5 [45.9 to 88.1]
  Length of chemotherapy cycle | 57.7 [36.2 to 76.5] | 47.7 [31.2 to 64.8]
  Medications taken | 48.2 [27.8 to 69.2] | 51.3 [34.4 to 67.9]
  Safety risk of intensive chemotherapy | 38.1 [20.5 to 59.6] | 25.9 [13.9 to 43.1]
  Planned relative dose intensity | 33.8 [20.3 to 50.7] | 30.7 [15.0 to 52.6]
  Patient lives far from clinic/healthcare resources | 29.9 [15.9 to 49.1] | 43.2 [28.2 to 59.5]
  Outpatient care of the patient | 22.5 [11.9 to 38.4] | 15.2 [7.1 to 29.6]
  Local access to reimbursed G-CSF PP | 21.2 [10.8 to 37.3] | 38.3 [19.8 to 61.0]
  Estimated compliance with the treatment plan | 19.9 [9.1 to 38.3] | 23.9 [13.3 to 39.1]
  Safety risk of G-CSFs in general | 18.7 [8.7 to 35.8] | 19.5 [7.8 to 40.9]
  Hospitalized patient | 17.6 [7.9 to 34.8] | 19.6 [10.1 to 34.4]
  Family/caregiver/nurse support to the patient | 14.5 [5.9 to 31.4] | 15.0 [6.5 to 31.1]
  Retired vs employed/active status of the patient | 8.5 [2.9 to 22.7] | 4.3 [1.0 to 16.9]
  Wait and see approach | 8.0 [2.8 to 20.9] | 15.2 [7.1 to 29.6]
  Private health insurance of the patient | 6.1 [1.8 to 18.1] | 8.4 [2.4 to 25.7]
  Other | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response. | 2.2 [0.3 to 15.3]

9. Secondary Outcome: Percentage of Participants for Whom Each Factor Was Ranked in the Granulocyte Colony Stimulating Factor (G-CSF) Primary Prophylaxis (PP) Decision as Important
Description: For each participant, the investigator ranked the factors that they considered to be the most important factors that they considered when deciding whether to use G-CSF PP treatment or not. To account for the expected correlation between participants with the same investigators and between investigators at the same sites, three-level, empty (no explanatory variables) multilevel models were used in the estimation of the percentages and 95% confidence intervals. ECOG = Eastern Cooperative Oncology Group.
Time Frame: At enrolment, prior to chemotherapy initiation.
Population: Primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Analysis Set
Number analyzed (Participants) | 944
percentage of participants
  Outcome of the overall FN risk assessment | 78.6 [71.4 to 84.3]
  Guidelines | 67.4 [53.4 to 78.9]
  Treatment intent | 67.1 [59.0 to 74.3]
  Age | 51.4 [42.9 to 59.8]
  ECOG/Karnofsky performance status | 36.1 [27.8 to 45.4]
  Baseline laboratory values | 18.1 [12.9 to 24.8]
  Length of chemotherapy cycle | 13.2 [8.5 to 20.1]
  Planned relative dose intensity | 9.6 [5.7 to 15.8]
  Outpatient care of the patient | 8.4 [5.3 to 13.1]
  Patient lives far from clinic/healthcare resources | 7.2 [4.7 to 11.0]
  Medications taken | 6.9 [4.4 to 10.5]
  Estimated compliance with the treatment plan | 4.8 [2.9 to 8.0]
  Safety risk of G-CSFs in general | 4.0 [2.5 to 6.1]
  Local access to reimbursed G-CSF PP | 3.4 [1.7 to 6.6]
  Family/caregiver/nurse support to the patient | 3.1 [1.8 to 5.3]
  Retired vs employed/active status of the patient | 3.1 [1.9 to 4.9]
  Hospitalized patient | 2.3 [1.3 to 4.0]
  Safety risk of intensive chemotherapy | 2.1 [1.2 to 3.6]
  Wait and see approach | 1.8 [1.0 to 3.3]
  Private health insurance of the patient | 1.0 [0.5 to 2.0]
  Other | 0.4 [0.1 to 1.2]

10. Secondary Outcome: Percentage of Participants for Whom Each Factor Was Ranked in the G-CSF PP Decision as Important by Country
Description: For each participant, the investigator ranked the risk factors that they considered to be the most important factors that they considered when deciding whether to use G-CSF PP treatment or not.
  To account for the expected correlation between participants with the same investigators and between investigators at the same sites, three-level, empty (no explanatory variables) multilevel models were used in the estimation of the percentages and 95% confidence intervals.
  ECOG = Eastern Cooperative Oncology Group.
Time Frame: At enrolment, prior to chemotherapy initiation.
Population: Primary analysis set; subgroup analyses were only performed on subgroups (countries) with at least 100 participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Poland | Greece | Romania | France
Number analyzed (Participants) | 205 | 173 | 141 | 126
percentage of participants
  Outcome of the overall FN risk assessment | 53.2 [30.4 to 74.7] | 60.3 [33.3 to 82.2] | 91.2 [82.4 to 95.8] | 74.5 [64.0 to 82.8]
  Guidelines | 79.9 [38.1 to 96.2] | 39.5 [13.8 to 72.7] | 87.2 [56.6 to 97.3] | 82.5 [40.1 to 97.1]
  Treatment intent | 62.6 [35.3 to 83.7] | 46.8 [27.9 to 66.7] | 81.0 [59.1 to 92.6] | 64.6 [42.3 to 81.9]
  Age | 59.9 [40.8 to 76.4] | 57.8 [36.2 to 76.8] | 54.2 [28.1 to 78.2] | 38.0 [20.9 to 58.6]
  ECOG/Karnofsky performance status | 69.3 [37.0 to 89.7] | 39.7 [20.7 to 62.5] | 34.6 [12.3 to 66.5] | 30.1 [18.4 to 45.1]
  Baseline laboratory values | 23.1 [11.3 to 41.5] | 9.7 [3.3 to 25.2] | 39.0 [20.9 to 60.7] | 4.3 [0.9 to 18.9]
  Length of chemotherapy cycle | 3.9 [1.7 to 8.4] | 20.0 [5.6 to 51.5] | 25.8 [8.2 to 57.4] | 5.6 [1.1 to 24.9]
  Planned relative dose intensity | 6.7 [2.8 to 15.4] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 11.3 [1.7 to 48.7] | 3.7 [0.8 to 15.9]
  Outpatient care of the patient | 3.5 [1.4 to 8.5] | 21.7 [6.0 to 54.4] | 10.9 [3.4 to 30.0] | 2.3 [0.3 to 14.9]
  Patient lives far from clinic/healthcare resources | 2.6 [1.0 to 6.2] | 14.3 [8.0 to 24.3] | 23.7 [10.7 to 44.5] | 3.5 [1.1 to 11.2]
  Medications taken | 3.7 [1.4 to 9.0] | 3.6 [1.0 to 11.9] | 8.0 [2.4 to 24.0] | 10.0 [4.2 to 22.0]
  Estimated compliance with the treatment plan | 1.2 [0.3 to 4.5] | 3.1 [0.6 to 15.2] | 8.6 [2.1 to 28.7] | 7.4 [1.5 to 30.0]
  Safety risk of G-CSFs in general | 5.0 [2.2 to 11.2] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response. | 2.1 [0.4 to 10.3]
  Local access to reimbursed G-CSF PP | 2.8 [0.7 to 10.0] | 1.4 [0.4 to 5.1] | 15.5 [2.9 to 52.8] | 1.0 [0.1 to 8.8]
  Family/caregiver/nurse support to the patient | 0.5 [0.1 to 3.6] | 3.4 [1.0 to 11.2] | 4.4 [1.3 to 13.8] | 4.4 [0.6 to 26.4]
  Retired vs employed/active status of the patient | 1.5 [0.5 to 4.7] | 5.3 [2.1 to 13.1] | 5.7 [1.7 to 17.6] | 2.5 [0.8 to 7.8]
  Hospitalized patient | 2.3 [0.8 to 6.4] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 5.0 [1.0 to 21.2] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model.
  Safety risk of intensive chemotherapy | 1.0 [0.3 to 4.0] | 1.2 [0.3 to 4.6] | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response. | 2.1 [0.4 to 9.9]
  Wait and see approach | 2.7 [0.9 to 7.9] | 4.4 [0.7 to 22.2] | 0.7 [0.1 to 5.0] | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response.
  Private health insurance of the patient | 1.4 [0.4 to 5.1] | 1.2 [0.3 to 4.6] | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response. | 0.8 [0.1 to 6.2]
  Other | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response. | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response. | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response. | 1.1 [0.1 to 9.5]

11. Secondary Outcome: Percentage of Participants for Whom Each Factor Was Ranked in the G-CSF PP Decision as Important by Clinical Specialty
Description: as for outcome 10
Time Frame: At enrolment, prior to chemotherapy initiation.
Population: Primary analysis set. Subgroup analyses were only performed in subgroups with at least 100 participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medical Oncologist | Hematologist
Number analyzed (Participants) | 662 | 140
percentage of participants
  Outcome of the overall FN risk assessment | 79.8 [71.5 to 86.1] | 78.6 [58.2 to 90.6]
  Guidelines | 72.6 [58.4 to 83.3] | 33.3 [12.8 to 63.0]
  Treatment intent | 69.9 [59.6 to 78.4] | 65.7 [50.8 to 78.1]
  Age | 50.2 [39.9 to 60.5] | 74.0 [61.8 to 83.3]
  ECOG/Karnofsky performance status | 37.6 [26.2 to 50.6] | 40.3 [29.1 to 52.6]
  Baseline laboratory values | 19.4 [13.3 to 27.5] | 25.2 [12.7 to 43.8]
  Length of chemotherapy cycle | 10.0 [5.9 to 16.4] | 24.0 [11.9 to 42.4]
  Planned relative dose intensity | 10.0 [5.5 to 17.5] | 18.8 [5.8 to 46.5]
  Outpatient care of the patient | 7.9 [4.5 to 13.4] | 16.1 [8.4 to 28.9]
  Patient lives far from clinic/healthcare resources | 9.0 [5.4 to 14.7] | 8.2 [3.8 to 16.9]
  Medications taken | 4.9 [3.0 to 8.0] | 17.9 [7.2 to 37.9]
  Estimated compliance with the treatment plan | 4.6 [2.3 to 8.9] | 8.6 [3.9 to 17.9]
  Safety risk of G-CSFs in general | 4.7 [3.0 to 7.4] | 4.2 [1.1 to 14.4]
  Local access to reimbursed G-CSF PP | 4.7 [2.1 to 10.2] | 4.2 [1.3 to 12.6]
  Family/caregiver/nurse support to the patient | 2.9 [1.6 to 5.2] | 5.5 [1.8 to 15.6]
  Retired vs employed/active status of the patient | 3.4 [1.9 to 5.9] | 4.7 [2.1 to 10.5]
  Hospitalized patient | 1.8 [0.9 to 3.6] | 5.9 [2.0 to 16.3]
  Safety risk of intensive chemotherapy | 2.3 [1.2 to 4.2] | 3.0 [1.0 to 8.9]
  Wait and see approach | 2.1 [1.1 to 3.9] | 3.8 [1.1 to 12.6]
  Private health insurance of the patient | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response.
  Other | 0.3 [0.1 to 1.4] | 1.0 [0.1 to 6.3]

12. Secondary Outcome: Percentage of Participants for Whom Each Factor Was Ranked in the G-CSF PP Decision as Important by Number of Years in Clinical Practice in Oncology / Hematology
Description: as for outcome 10
Time Frame: At enrolment, prior to chemotherapy initiation.
Population: Primary analysis set. Subgroup analyses were only performed in subgroups with at least 100 participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ≤ 10 Years | > 10 Years
Number analyzed (Participants) | 257 | 687
percentage of participants
  Outcome of the overall FN risk assessment | 76.6 [60.4 to 87.5] | 76.8 [69.7 to 82.7]
  Guidelines | 59.3 [35.9 to 79.2] | 65.2 [50.5 to 77.5]
  Treatment intent | 57.7 [42.9 to 71.1] | 71.1 [62.0 to 78.8]
  Age | 55.2 [38.5 to 70.8] | 50.2 [41.7 to 58.8]
  ECOG/Karnofsky performance status | 28.8 [18.0 to 42.6] | 40.2 [30.9 to 50.3]
  Baseline laboratory values | 14.9 [8.7 to 24.3] | 18.6 [12.8 to 26.0]
  Length of chemotherapy cycle | 16.6 [8.6 to 29.6] | 12.5 [7.6 to 20.0]
  Planned relative dose intensity | 7.9 [3.4 to 17.1] | 9.5 [5.2 to 16.8]
  Outpatient care of the patient | 10.2 [4.9 to 19.8] | 8.5 [5.1 to 13.7]
  Patient lives far from clinic/healthcare resources | 5.3 [2.4 to 11.2] | 8.3 [5.3 to 12.7]
  Medications taken | 4.3 [2.1 to 8.8] | 7.6 [4.7 to 12.1]
  Estimated compliance with the treatment plan | 4.0 [1.6 to 9.7] | 5.4 [3.1 to 9.1]
  Safety risk of G-CSFs in general | 3.4 [1.5 to 7.6] | 4.0 [2.3 to 6.7]
  Local access to reimbursed G-CSF PP | 3.9 [1.4 to 10.3] | 3.6 [1.7 to 7.4]
  Family/caregiver/nurse support to the patient | 6.2 [3.0 to 12.5] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model.
  Retired vs employed/active status of the patient | 3.5 [1.6 to 7.4] | 3.1 [1.8 to 5.3]
  Hospitalized patient | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 2.6 [1.3 to 5.1]
  Safety risk of intensive chemotherapy | 1.8 [0.6 to 5.0] | 2.4 [1.4 to 4.2]
  Wait and see approach | 1.5 [0.5 to 4.7] | 2.0 [1.0 to 3.9]
  Private health insurance of the patient | 0.4 [0.1 to 2.9] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model.
  Other | 0.4 [0.1 to 2.8] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model.

13. Secondary Outcome: Percentage of Participants for Whom Each Factor Was Ranked in the G-CSF PP Decision as Important by Institution Type
Description: as for outcome 10
Time Frame: At enrolment, prior to chemotherapy initiation.
Population: Primary analysis set. Subgroup analyses were only performed in subgroups with at least 100 participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | University Hospital | General Hospital | Private Center | Comprehensive Cancer Center
Number analyzed (Participants) | 302 | 281 | 197 | 164
percentage of participants
  Outcome of the overall FN risk assessment | 78.1 [65.5 to 87.0] | 73.4 [56.3 to 85.5] | 90.6 [80.8 to 95.7] | 62.4 [39.8 to 80.7]
  Guidelines | 68.2 [38.6 to 88.0] | 65.2 [46.5 to 80.1] | 82.3 [57.1 to 94.2] | 41.8 [10.1 to 82.2]
  Treatment intent | 71.7 [58.2 to 82.2] | 67.3 [52.9 to 79.0] | 63.5 [42.5 to 80.3] | 62.0 [39.4 to 80.4]
  Age | 41.1 [27.7 to 56.0] | 58.4 [41.3 to 73.7] | 52.6 [36.9 to 67.8] | 67.3 [50.3 to 80.7]
  ECOG/Karnofsky performance status | 29.3 [18.8 to 42.6] | 39.1 [26.0 to 54.0] | 35.2 [17.8 to 57.7] | 53.3 [23.3 to 81.1]
  Baseline laboratory values | 18.9 [10.2 to 32.2] | 16.1 [8.0 to 29.7] | 13.5 [5.7 to 28.6] | 29.9 [15.5 to 49.6]
  Length of chemotherapy cycle | 26.5 [12.4 to 48.0] | 13.4 [7.9 to 21.9] | 4.8 [1.6 to 13.2] | 7.8 [3.2 to 17.5]
  Planned relative dose intensity | 13.1 [4.5 to 32.4] | 7.0 [2.6 to 17.6] | 8.8 [3.2 to 21.7] | 8.1 [2.1 to 26.7]
  Outpatient care of the patient | 5.4 [2.0 to 14.3] | 11.5 [6.3 to 20.2] | 11.9 [4.5 to 27.7] | 4.0 [1.0 to 14.2]
  Patient lives far from clinic/healthcare resources | 6.6 [2.4 to 16.8] | 11.6 [7.3 to 18.0] | 6.1 [2.5 to 14.5] | 2.5 [0.6 to 9.2]
  Medications taken | 7.4 [3.2 to 16.2] | 7.9 [3.5 to 16.8] | 5.0 [2.0 to 11.8] | 6.1 [1.4 to 23.4]
  Estimated compliance with the treatment plan | 5.2 [2.0 to 12.5] | 4.6 [1.9 to 10.5] | 5.2 [1.6 to 15.6] | 3.0 [0.6 to 14.2]
  Safety risk of G-CSFs in general | 2.7 [1.2 to 6.1] | 5.2 [2.7 to 9.6] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 9.7 [3.5 to 24.1]
  Local access to reimbursed G-CSF PP | 1.9 [0.4 to 7.7] | 9.0 [3.6 to 20.6] | 2.1 [0.4 to 11.6] | 1.7 [0.4 to 8.0]
  Family/caregiver/nurse support to the patient | 3.3 [1.4 to 7.6] | 3.2 [1.2 to 8.3] | 2.9 [0.8 to 10.8] | 1.6 [0.3 to 9.6]
  Retired vs employed/active status of the patient | 2.9 [1.3 to 6.5] | 3.8 [1.6 to 8.8] | 3.0 [1.2 to 7.2] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model.
  Hospitalized patient | 2.8 [1.0 to 8.2] | 1.9 [0.6 to 5.6] | 2.3 [0.7 to 7.0] | 1.3 [0.3 to 5.1]
  Safety risk of intensive chemotherapy | 1.8 [0.6 to 5.2] | 2.3 [0.9 to 6.1] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 3.4 [1.1 to 9.8]
  Wait and see approach | 0.7 [0.2 to 2.6] | 1.3 [0.4 to 4.5] | 2.8 [0.8 to 9.5] | 3.5 [0.8 to 14.5]
  Private health insurance of the patient | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response. | 1.7 [0.6 to 4.8] | 1.4 [0.4 to 4.6] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model.
  Other | 0.9 [0.2 to 3.8] | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response. | 0.5 [0.1 to 3.6] | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response.

14. Secondary Outcome: Percentage of Participants for Whom Each Factor Was Ranked in the G-CSF PP Decision as Important by Tumor Type
Description: as for outcome 10
Time Frame: At enrolment, prior to chemotherapy initiation.
Population: Primary analysis set. Subgroup analyses were only performed in subgroups with at least 100 participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Breast Cancer | Non-small Cell Lung Cancer | Non-Hodgkin's Lymphoma | Small Cell Lung Cancer
Number analyzed (Participants) | 395 | 248 | 182 | 119
percentage of participants
  Outcome of the overall FN risk assessment | 81.4 [73.9 to 87.2] | 64.5 [51.4 to 75.8] | 78.5 [64.1 to 88.2] | 62.6 [47.2 to 75.8]
  Guidelines | 75.5 [62.3 to 85.1] | 59.7 [39.5 to 77.0] | 45.4 [25.1 to 67.4] | 59.8 [35.7 to 79.9]
  Treatment intent | 68.8 [57.1 to 78.6] | 66.6 [56.4 to 75.4] | 60.5 [46.9 to 72.6] | 62.7 [48.2 to 75.2]
  Age | 39.1 [28.9 to 50.2] | 56.5 [44.1 to 68.1] | 69.5 [57.7 to 79.2] | 45.1 [30.7 to 60.4]
  ECOG/Karnofsky performance status | 25.9 [17.3 to 36.9] | 49.5 [34.3 to 64.7] | 42.1 [30.0 to 55.2] | 44.0 [28.3 to 60.9]
  Baseline laboratory values | 16.3 [11.3 to 22.8] | 24.2 [15.4 to 35.9] | 29.1 [18.7 to 42.3] | 9.7 [4.0 to 21.5]
  Length of chemotherapy cycle | 10.4 [5.8 to 17.9] | 16.1 [7.8 to 30.1] | 16.7 [8.4 to 30.4] | 14.5 [6.2 to 30.3]
  Planned relative dose intensity | 9.1 [4.5 to 17.3] | 7.2 [3.5 to 14.1] | 18.1 [7.5 to 37.7] | 13.1 [6.7 to 24.0]
  Outpatient care of the patient | 7.7 [4.1 to 14.0] | 12.7 [6.3 to 23.7] | 10.3 [5.1 to 19.9] | 10.4 [3.6 to 26.6]
  Patient lives far from clinic/healthcare resources | 7.6 [4.1 to 13.9] | 8.9 [4.7 to 16.4] | 8.2 [4.2 to 15.4] | 5.8 [2.3 to 13.8]
  Medications taken | 3.9 [1.9 to 7.9] | 4.1 [1.9 to 8.4] | 15.0 [7.1 to 29.1] | 7.9 [4.1 to 14.6]
  Estimated compliance with the treatment plan | 5.1 [2.5 to 10.1] | 4.3 [1.7 to 10.5] | 7.2 [3.3 to 15.3] | 5.0 [1.7 to 13.7]
  Safety risk of G-CSFs in general | 5.0 [2.9 to 8.5] | 2.7 [1.2 to 6.0] | 5.4 [2.1 to 13.1] | 5.2 [2.1 to 12.4]
  Local access to reimbursed G-CSF PP | 5.0 [2.1 to 11.2] | 6.9 [2.6 to 16.6] | 5.7 [2.3 to 13.4] | 7.4 [2.6 to 18.9]
  Family/caregiver/nurse support to the patient | 2.7 [1.2 to 5.9] | 3.3 [1.6 to 6.8] | 4.5 [1.8 to 11.0] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model.
  Retired vs employed/active status of the patient | 3.2 [1.6 to 6.1] | 2.6 [1.1 to 6.1] | 4.1 [1.9 to 8.4] | 3.9 [1.2 to 11.7]
  Hospitalized patient | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 4.2 [2.0 to 8.5] | 4.9 [1.9 to 12.0] | 1.8 [0.4 to 7.7]
  Safety risk of intensive chemotherapy | 2.7 [1.3 to 5.3] | 0.8 [0.2 to 3.3] | 3.5 [1.5 to 8.2] | 2.6 [0.8 to 8.0]
  Wait and see approach | 2.3 [1.1 to 4.8] | 3.2 [1.3 to 7.4] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 2.9 [0.9 to 9.2]
  Private health insurance of the patient | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 2.1 [0.8 to 5.6] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 1.8 [0.4 to 7.3]
  Other | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 0.7 [0.1 to 4.5] | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response.

15. Secondary Outcome: Percentage of Investigators Who Ranked Each Factor as a Risk Factor for Febrile Neutropenia by Clinical Specialty
Description: During the baseline investigator assessment (prior to identification of participants), investigators were provided a list of risk factors on a source document worksheet, and asked to rankt the risk factors that they considered to be the most important when assessing overall FN risk. To account for the expected correlation between investigators at the same sites, two-level, empty (no explanatory variables) multilevel models were used in the estimation of the percentages and 95% confidence intervals. ECOG = Eastern Cooperative Oncology Group. Subgroup analyses were performed where a subgroup contained at least 40 investigators. Results are reported for medical oncologists as this was the only specialty that contained at least 40 investigators.
Time Frame: Assessed at Baseline, prior to participant enrolment.
Population: Primary analysis set - investigators (PASI); analysis was only performed for subgroups containing at least 40 investigators.
Measure: Number (95% Confidence Interval); unit: percentage of investigators
Units Other Than Participants: Investigators
Arm/Group | Medical Oncologist
Number analyzed (Participants) | 662
Number analyzed (Investigators) | 110
percentage of investigators
  Chemotherapy agents in the backbone | 88.5 [80.6 to 93.5]
  History of prior FN | 82.2 [73.2 to 88.6]
  Guidelines | 74.7 [62.8 to 83.8]
  Baseline laboratory values | 71.4 [61.3 to 79.7]
  Age | 68.6 [58.3 to 77.3]
  Prior chemotherapy | 67.4 [57.6 to 75.8]
  ECOG/Karnofsky performance status | 64.6 [53.7 to 74.1]
  Comorbidities | 64.4 [53.8 to 73.7]
  Tumor stage | 64.3 [53.6 to 73.8]
  Prior radiotherapy involving bone marrow | 63.3 [52.7 to 72.7]
  Documented bone marrow involvement | 57.3 [44.4 to 69.4]
  Tumor type | 56.5 [45.1 to 67.2]
  Treatment intent | 55.0 [44.1 to 65.5]
  Nutritional status | 53.6 [41.8 to 65.0]
  Medications taken | 49.4 [37.8 to 61.2]
  Current infection | 44.8 [34.0 to 56.1]
  Open wounds | 42.4 [29.8 to 56.1]
  Personal experience of chemotherapy regimen risk | 40.9 [31.5 to 51.1]
  Concurrent radiotherapy | 39.7 [27.6 to 53.1]
  Female gender | 32.4 [21.1 to 46.0]
  Planned relative dose intensity | 29.6 [20.5 to 40.8]
  Other disease/treatment related | 5.4 [2.2 to 12.3]
  Other patient related | 2.7 [0.9 to 8.3]

16. Secondary Outcome: Percentage of Investigators Who Ranked Each Factor as a Risk Factor for Febrile Neutropenia by Number of Years in Clinical Practice in Oncology / Hematology
Description: During the baseline investigator assessment (prior to identification of participants), investigators were provided a list of risk factors on a source document worksheet, and asked to rank the risk factors that they considered to be the most important when assessing overall FN risk. To account for the expected correlation between investigators at the same sites, two-level, empty (no explanatory variables) multilevel models were used in the estimation of the percentages and 95% confidence intervals. ECOG = Eastern Cooperative Oncology Group.
Time Frame: Assessed at Baseline, prior to participant enrolment.
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of investigators
Units Other Than Participants: Investigators
Arm/Group | ≤ 10 Years | > 10 Years
Number analyzed (Participants) | 257 | 687
Number analyzed (Investigators) | 48 | 117
percentage of investigators
  Chemotherapy agents in the backbone | 89.6 [75.6 to 96.0] | 87.4 [79.3 to 92.7]
  History of prior FN | 89.5 [74.5 to 96.1] | 79.6 [70.9 to 86.2]
  Guidelines | 73.1 [57.0 to 84.7] | 67.3 [56.1 to 76.8]
  Baseline laboratory values | 71.5 [54.8 to 83.8] | 76.1 [67.3 to 83.2]
  Age | 68.9 [52.8 to 81.4] | 74.9 [64.3 to 83.2]
  Prior chemotherapy | 68.8 [52.3 to 81.7] | 71.1 [61.7 to 78.9]
  ECOG/Karnofsky performance status | 54.9 [37.4 to 71.2] | 68.1 [57.4 to 77.1]
  Comorbidities | 52.1 [36.8 to 67.0] | 67.0 [57.0 to 75.7]
  Tumor stage | 60.9 [43.4 to 76.0] | 61.5 [51.3 to 70.8]
  Prior radiotherapy involving bone marrow | 65.0 [47.3 to 79.3] | 63.8 [53.9 to 72.6]
  Documented bone marrow involvement | 58.6 [41.5 to 73.9] | 62.7 [50.9 to 73.2]
  Tumor type | 60.8 [44.2 to 75.2] | 63.4 [52.5 to 73.0]
  Treatment intent | 47.9 [33.0 to 63.2] | 52.2 [41.0 to 63.3]
  Nutritional status | 46.7 [28.1 to 66.4] | 49.3 [39.7 to 58.9]
  Medications taken | 45.3 [26.7 to 65.3] | 48.8 [38.2 to 59.5]
  Current infection | 39.6 [24.7 to 56.7] | 47.3 [37.5 to 57.3]
  Open wounds | 30.1 [16.7 to 48.1] | 40.5 [29.9 to 52.0]
  Personal experience of chemotherapy regimen risk | 33.3 [20.5 to 49.2] | 43.5 [34.4 to 53.1]
  Concurrent radiotherapy | 44.0 [27.8 to 61.6] | 41.4 [31.3 to 52.3]
  Female gender | 22.9 [11.9 to 39.5] | 24.5 [16.3 to 35.1]
  Planned relative dose intensity | 27.1 [15.6 to 42.8] | 25.8 [17.8 to 35.8]
  Other disease/treatment related | 4.8 [1.1 to 19.0] | 3.8 [1.4 to 9.6]
  Other patient related | 2.1 [0.2 to 15.9] | 2.6 [0.8 to 7.9]

17. Secondary Outcome: Percentage of Investigators Who Ranked Each Factor as a Risk Factor for Febrile Neutropenia by Institution Type
Description: During the baseline investigator assessment (prior to identification of participants), investigators were provided a list of risk factors on a source document worksheet, and asked to rank the factors that they considered to be the most important when assessing overall FN risk. To account for the expected correlation between investigators at the same sites, two-level, empty (no explanatory variables) multilevel models were used in the estimation of the percentages and 95% confidence intervals. ECOG = Eastern Cooperative Oncology Group.
Time Frame: Assessed at Baseline, prior to participant enrolment.
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of investigators
Units Other Than Participants: Investigators
Arm/Group | University Hospital | General Hospital
Number analyzed (Participants) | 302 | 281
Number analyzed (Investigators) | 57 | 46
percentage of investigators
  Chemotherapy agents in the backbone | 91.2 [75.6 to 97.2] | 87.0 [72.9 to 94.3]
  History of prior FN | 87.5 [73.3 to 94.7] | 78.3 [61.1 to 89.3]
  Guidelines | 73.1 [54.1 to 86.2] | 62.9 [45.4 to 77.6]
  Baseline laboratory values | 83.1 [64.8 to 92.9] | 79.4 [63.0 to 89.7]
  Age | 72.5 [53.5 to 85.7] | 77.2 [55.9 to 90.0]
  Prior chemotherapy | 75.1 [57.3 to 87.1] | 72.0 [53.0 to 85.4]
  ECOG/Karnofsky performance status | 58.4 [42.3 to 72.9] | 74.1 [57.4 to 85.9]
  Comorbidities | 68.4 [54.7 to 79.5] | 62.0 [41.1 to 79.3]
  Tumor stage | 58.6 [38.1 to 76.5] | 64.5 [47.3 to 78.6]
  Prior radiotherapy involving bone marrow | 76.8 [57.9 to 88.8] | 61.5 [41.2 to 78.5]
  Documented bone marrow involvement | 78.3 [58.7 to 90.2] | 63.0 [44.0 to 78.6]
  Tumor type | 65.3 [44.8 to 81.4] | 60.9 [45.4 to 74.4]
  Treatment intent | 49.6 [30.9 to 68.4] | 47.8 [33.2 to 62.8]
  Nutritional status | 46.7 [30.9 to 63.1] | 47.0 [26.7 to 68.2]
  Medications taken | 51.5 [31.1 to 71.3] | 50.8 [34.7 to 66.7]
  Current infection | 40.7 [26.0 to 57.3] | 55.6 [37.9 to 71.9]
  Open wounds | 44.6 [29.5 to 60.9] | 39.0 [20.8 to 60.9]
  Personal experience of chemotherapy regimen risk | 32.6 [19.6 to 49.0] | 39.0 [23.7 to 56.9]
  Concurrent radiotherapy | 45.9 [29.1 to 63.8] | 34.2 [18.0 to 55.2]
  Female gender | 19.2 [9.5 to 35.0] | 10.2 [3.1 to 28.4]
  Planned relative dose intensity | 21.7 [11.2 to 37.8] | 23.1 [10.7 to 43.0]
  Other disease/treatment related | 3.5 [0.8 to 14.6] | 2.6 [0.3 to 17.4]
  Other patient related | 3.5 [0.8 to 14.1] | 2.2 [0.3 to 15.3]

18. Secondary Outcome: Percentage of Participants for Whom Each FN Risk Factor Was Ranked as Important by Country
Description: as for outcome 4
Time Frame: At enrolment, prior to chemotherapy initiation.
Population: Primary analysis set; analysis only includes subgroups with at least 100 participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Poland | Greece | Romania | France
Number analyzed (Participants) | 205 | 173 | 141 | 126
percentage of participants
  Chemotherapy agents in the backbone | 81.4 [49.6 to 95.1] | 96.3 [80.7 to 99.4] | 98.2 [90.4 to 99.7] | 88.3 [59.0 to 97.5]
  Tumor type | 67.8 [28.1 to 91.9] | 61.4 [18.3 to 91.8] | 95.3 [82.6 to 98.9] | 67.9 [44.2 to 85.0]
  Guidelines | 85.3 [40.9 to 98.0] | 44.7 [21.4 to 70.6] | 91.0 [62.9 to 98.4] | 62.7 [24.1 to 89.9]
  Tumor stage | 47.3 [14.3 to 82.8] | 39.5 [17.9 to 66.0] | 69.4 [45.6 to 86.0] | 24.3 [11.4 to 44.3]
  Age | 50.1 [27.8 to 72.4] | 45.1 [24.7 to 67.3] | 33.0 [19.6 to 50.0] | 13.5 [5.2 to 30.8]
  Treatment intent | 15.8 [6.5 to 33.7] | 24.7 [12.2 to 43.5] | 52.0 [33.0 to 70.4] | 16.9 [3.9 to 50.1]
  ECOG/Karnofsky performance status | 57.4 [29.8 to 81.1] | 29.3 [15.2 to 48.9] | 23.4 [8.0 to 51.9] | 19.4 [10.6 to 32.9]
  Female gender | 28.9 [15.0 to 48.3] | 4.1 [1.1 to 13.7] | 38.0 [18.3 to 62.6] | 8.7 [2.8 to 24.1]
  Comorbidities | 18.3 [11.7 to 27.5] | 18.2 [11.7 to 27.1] | 29.9 [14.5 to 51.9] | 6.4 [2.0 to 18.2]
  Baseline laboratory values | 18.5 [10.1 to 31.4] | 7.9 [2.3 to 23.3] | 27.7 [11.1 to 54.1] | 7.4 [2.4 to 20.6]
  Personal experience of chemotherapy regimen risk | 4.5 [1.1 to 16.7] | 19.2 [6.4 to 45.1] | 11.6 [2.9 to 36.7] | 26.8 [15.0 to 43.2]
  Prior chemotherapy | 14.1 [8.2 to 23.4] | 12.7 [7.1 to 21.7] | 28.8 [15.0 to 48.2] | 10.7 [5.4 to 20.2]
  Nutritional status | 9.0 [4.3 to 18.0] | 2.6 [0.5 to 11.6] | 12.6 [4.9 to 28.7] | 10.7 [4.9 to 21.6]
  Planned relative dose intensity | 4.3 [1.4 to 12.5] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 12.0 [1.4 to 57.1] | 3.5 [0.9 to 12.4]
  Medications taken | 1.9 [0.6 to 5.8] | 4.2 [1.7 to 10.0] | 5.0 [1.8 to 13.0] | 4.2 [1.5 to 11.5]
  History of prior FN | 4.4 [1.2 to 15.2] | 2.9 [1.2 to 6.8] | 7.3 [3.2 to 15.9] | 4.0 [1.2 to 13.1]
  Documented bone marrow involvement | 1.0 [0.2 to 3.8] | 8.0 [2.1 to 26.3] | 2.6 [0.6 to 10.5] | 2.1 [0.5 to 8.7]
  Prior radiotherapy involving bone marrow | 5.2 [2.5 to 10.6] | 3.6 [1.2 to 10.2] | 3.1 [1.0 to 9.3] | 1.6 [0.4 to 6.6]
  Current infection | 2.9 [1.2 to 6.7] | 4.0 [1.9 to 8.5] | 3.1 [0.6 to 15.0] | 1.0 [0.1 to 7.4]
  Concurrent radiotherapy | 2.3 [0.9 to 5.9] | 5.7 [2.2 to 13.6] | 0.7 [0.1 to 5.4] | 3.5 [1.0 to 11.0]
  Open wounds | 1.7 [0.5 to 5.4] | 0.7 [0.1 to 4.3] | 1.7 [0.4 to 6.5] | 0.8 [0.1 to 6.3]
  Other patient related | 0.5 [0.1 to 3.6] | 1.9 [0.4 to 9.0] | 2.5 [0.8 to 7.8] | 1.2 [0.2 to 6.0]
  Other disease/treatment related | 2.3 [0.8 to 6.5] | 0.6 [0.1 to 4.2] | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response. | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response.

19. Secondary Outcome: Percentage of Participants for Whom Each FN Risk Factor Was Ranked as Important by Clinical Specialty
Description: as for outcome 4
Time Frame: At enrolment, prior to chemotherapy initiation.
Population: Primary analysis set; analysis only included subgroups with at least 100 participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medical Oncologist | Hematologist
Number analyzed (Participants) | 662 | 140
percentage of participants
  Chemotherapy agents in the backbone | 93.1 [87.5 to 96.3] | 93.6 [84.4 to 97.5]
  Tumor type | 72.6 [59.0 to 83.0] | 81.4 [59.4 to 92.9]
  Guidelines | 71.9 [58.0 to 82.6] | 27.5 [11.0 to 53.7]
  Tumor stage | 49.0 [37.8 to 60.3] | 42.3 [26.3 to 60.2]
  Age | 40.9 [32.4 to 50.1] | 55.5 [42.2 to 68.0]
  Treatment intent | 30.4 [22.5 to 39.7] | 39.0 [23.7 to 56.8]
  ECOG/Karnofsky performance status | 30.2 [21.1 to 41.1] | 28.8 [18.8 to 41.6]
  Female gender | 22.2 [14.6 to 32.3] | 13.6 [8.0 to 22.1]
  Comorbidities | 13.8 [10.2 to 18.3] | 27.2 [17.2 to 40.2]
  Baseline laboratory values | 15.1 [10.5 to 21.3] | 24.7 [14.2 to 39.5]
  Personal experience of chemotherapy regimen risk | 17.3 [10.4 to 27.5] | 10.0 [4.5 to 20.8]
  Prior chemotherapy | 15.7 [11.3 to 21.3] | 14.4 [9.2 to 21.8]
  Nutritional status | 7.3 [4.7 to 11.1] | 13.2 [6.7 to 24.5]
  Planned relative dose intensity | 7.8 [4.0 to 14.6] | 9.4 [3.1 to 24.9]
  Medications taken | 4.0 [2.6 to 6.3] | 11.9 [5.6 to 23.4]
  History of prior FN | 3.6 [2.1 to 6.1] | 5.7 [2.5 to 12.6]
  Documented bone marrow involvement | 2.1 [1.2 to 3.7] | 20.8 [12.2 to 33.1]
  Prior radiotherapy involving bone marrow | 4.4 [3.0 to 6.5] | 2.9 [1.1 to 7.4]
  Current infection | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 9.1 [4.3 to 18.3]
  Concurrent radiotherapy | 2.3 [1.4 to 4.0] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model.
  Open wounds | 2.4 [1.3 to 4.4] | 2.7 [0.8 to 8.5]
  Other patient related | 1.3 [0.6 to 2.9] | 4.4 [1.6 to 11.7]
  Other disease/treatment related | 1.2 [0.5 to 2.6] | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response.

20. Secondary Outcome: Percentage of Participants for Whom Each FN Risk Factor Was Ranked as Important by Number of Years in Clinical Practice in Oncology / Hematology
Description: as for outcome 4
Time Frame: At enrolment, prior to chemotherapy initiation.
Population: Primary analysis set; analysis only included subgroups with at least 100 participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ≤ 10 Years | > 10 Years
Number analyzed (Participants) | 257 | 687
percentage of participants
  Chemotherapy agents in the backbone | 91.5 [80.2 to 96.6] | 92.6 [87.5 to 95.7]
  Tumor type | 59.1 [41.0 to 75.0] | 76.6 [65.0 to 85.3]
  Guidelines | 55.7 [32.8 to 76.5] | 60.1 [45.9 to 72.8]
  Tumor stage | 34.9 [22.6 to 49.6] | 45.9 [35.3 to 56.8]
  Age | 35.5 [24.1 to 48.9] | 41.5 [33.3 to 50.2]
  Treatment intent | 26.8 [17.7 to 38.3] | 32.3 [23.8 to 42.2]
  ECOG/Karnofsky performance status | 23.5 [14.1 to 36.3] | 31.1 [23.8 to 39.6]
  Female gender | 12.5 [7.6 to 20.0] | 21.1 [14.1 to 30.2]
  Comorbidities | 14.7 [9.9 to 21.4] | 16.2 [12.4 to 20.8]
  Baseline laboratory values | 12.6 [7.0 to 21.7] | 15.5 [11.0 to 21.3]
  Personal experience of chemotherapy regimen risk | 15.8 [8.2 to 28.3] | 15.1 [9.7 to 22.7]
  Prior chemotherapy | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 15.8 [11.9 to 20.6]
  Nutritional status | 5.3 [2.5 to 11.0] | 9.2 [6.5 to 12.9]
  Planned relative dose intensity | 5.1 [2.2 to 11.7] | 7.7 [4.3 to 13.6]
  Medications taken | 5.3 [3.0 to 9.5] | 5.0 [3.1 to 7.9]
  History of prior FN | 2.2 [0.8 to 5.4] | 5.1 [3.3 to 7.9]
  Documented bone marrow involvement | 3.2 [1.5 to 6.7] | 4.8 [2.8 to 8.2]
  Prior radiotherapy involving bone marrow | 3.9 [2.1 to 7.1] | 4.1 [2.8 to 6.2]
  Current infection | 1.8 [0.7 to 4.7] | 4.5 [2.8 to 7.1]
  Concurrent radiotherapy | 3.8 [1.8 to 8.0] | 2.1 [1.2 to 3.7]
  Open wounds | 0.9 [0.2 to 3.3] | 2.7 [1.5 to 4.8]
  Other patient related | 2.8 [1.1 to 6.6] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model.
  Other disease/treatment related | 1.5 [0.5 to 4.5] | 0.5 [0.2 to 1.5]

21. Secondary Outcome: Percentage of Participants for Whom Each FN Risk Factor Was Ranked as Important by Institution Type
Description: as for outcome 4
Time Frame: At enrolment, prior to chemotherapy initiation.
Population: Primary analysis set; analysis only included subgroups with at least 100 participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | University Hospital | General Hospital | Private Center | Comprehensive Cancer Center
Number analyzed (Participants) | 302 | 281 | 197 | 164
percentage of participants
  Chemotherapy agents in the backbone | 95.4 [87.7 to 98.4] | 92.7 [83.1 to 97.0] | 91.9 [76.1 to 97.6] | 86.1 [68.3 to 94.6]
  Tumor type | 66.2 [44.8 to 82.5] | 81.6 [60.1 to 92.9] | 68.7 [42.0 to 86.9] | 74.4 [38.9 to 93.0]
  Guidelines | 51.5 [27.6 to 74.8] | 64.0 [46.5 to 78.5] | 74.8 [46.8 to 90.9] | 54.6 [12.0 to 91.4]
  Tumor stage | 37.3 [21.7 to 56.0] | 51.4 [38.7 to 63.9] | 36.9 [20.4 to 57.2] | 44.8 [16.3 to 77.3]
  Age | 33.5 [20.1 to 50.2] | 37.8 [25.6 to 51.9] | 45.8 [31.5 to 60.9] | 50.3 [29.9 to 70.6]
  Treatment intent | 32.0 [19.0 to 48.4] | 33.7 [21.1 to 49.0] | 33.1 [19.9 to 49.5] | 17.2 [8.0 to 33.1]
  ECOG/Karnofsky performance status | 20.6 [12.9 to 31.2] | 31.7 [19.9 to 46.4] | 29.3 [15.2 to 49.1] | 42.1 [21.5 to 65.9]
  Female gender | 14.9 [7.4 to 27.9] | 15.8 [8.2 to 28.4] | 22.6 [9.7 to 44.4] | 25.4 [12.1 to 45.7]
  Comorbidities | 14.3 [8.6 to 22.9] | 13.9 [9.3 to 20.1] | 17.8 [9.8 to 30.1] | 17.3 [10.6 to 27.0]
  Baseline laboratory values | 20.5 [10.5 to 36.2] | 12.5 [7.4 to 20.4] | 10.5 [4.4 to 23.0] | 22.1 [12.9 to 35.2]
  Personal experience of chemotherapy regimen risk | 9.4 [4.4 to 19.0] | 15.4 [7.6 to 28.6] | 37.6 [22.2 to 55.9] | 4.8 [1.5 to 14.5]
  Prior chemotherapy | 15.9 [9.5 to 25.3] | 13.0 [9.2 to 18.0] | 12.8 [7.0 to 22.4] | 18.5 [6.5 to 42.4]
  Nutritional status | 8.3 [4.2 to 15.8] | 11.2 [6.2 to 19.4] | 5.4 [2.4 to 11.6] | 5.9 [2.6 to 12.8]
  Planned relative dose intensity | 10.5 [3.9 to 25.1] | 6.3 [2.4 to 15.5] | 4.1 [1.0 to 15.4] | 7.7 [1.9 to 26.5]
  Medications taken | 6.2 [3.2 to 11.5] | 7.3 [3.5 to 14.6] | 2.9 [1.2 to 7.0] | 3.2 [0.9 to 10.5]
  History of prior FN | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 3.0 [1.3 to 6.5] | 5.6 [2.7 to 11.3] | 3.9 [0.9 to 16.0]
  Documented bone marrow involvement | 6.4 [2.9 to 13.8] | 5.0 [2.3 to 10.7] | 3.6 [1.2 to 10.5] | 0.6 [0.1 to 4.4]
  Prior radiotherapy involving bone marrow | 3.1 [1.4 to 6.9] | 2.8 [1.4 to 5.6] | 5.2 [2.6 to 10.0] | 4.4 [1.9 to 9.9]
  Current infection | 4.9 [2.1 to 10.8] | 2.9 [1.2 to 6.8] | 3.3 [1.1 to 9.3] | 2.9 [1.1 to 7.7]
  Concurrent radiotherapy | 1.4 [0.5 to 4.3] | 2.1 [0.8 to 5.4] | 3.1 [1.3 to 7.3] | 2.2 [0.9 to 6.4]
  Open wounds | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 1.8 [0.6 to 5.4] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 3.0 [1.1 to 7.8]
  Other patient related | 3.6 [1.4 to 9.1] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 2.4 [0.9 to 6.6] | 1.2 [0.3 to 5.1]
  Other disease/treatment related | 0 [NA to NA] — Not applicable since the statistical model was not applied to calculate confidence limits for outcomes with no variation in response. | 1.3 [0.5 to 3.8] | 0.6 [0.1 to 4.8] | 1.7 [0.5 to 5.9]

22. Secondary Outcome: Percentage of Participants for Whom Each FN Risk Factor Was Ranked as Important by Tumor Type
Description: as for outcome 4
Time Frame: At enrolment, prior to chemotherapy initiation.
Population: Primary analysis set; analysis only included subgroups with at least 100 participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Breast Cancer | Non-small Cell Lung Cancer | Non-Hodgkin's Lymphoma | Small Cell Lung Cancer
Number analyzed (Participants) | 395 | 248 | 182 | 119
percentage of participants
  Chemotherapy agents in the backbone | 93.8 [88.9 to 96.6] | 85.8 [71.6 to 93.5] | 90.6 [81.8 to 95.4] | 80.5 [62.0 to 91.2]
  Tumor type | 64.9 [49.4 to 77.8] | 75.9 [58.2 to 87.7] | 77.4 [59.6 to 88.8] | 64.7 [50.2 to 76.9]
  Guidelines | 68.4 [55.5 to 78.9] | 62.7 [43.2 to 78.8] | 43.2 [23.2 to 65.7] | 56.3 [33.4 to 76.7]
  Tumor stage | 38.7 [28.3 to 50.2] | 57.7 [42.1 to 72.0] | 39.7 [26.6 to 54.4] | 64.7 [36.7 to 71.5]
  Age | 31.7 [23.5 to 41.3] | 42.3 [30.3 to 55.3] | 56.9 [45.9 to 67.2] | 33.5 [19.3 to 51.6]
  Treatment intent | 34.0 [23.9 to 45.7] | 25.2 [16.4 to 36.7] | 35.1 [23.4 to 48.9] | 22.2 [11.8 to 37.9]
  ECOG/Karnofsky performance status | 21.1 [13.8 to 30.8] | 40.7 [27.8 to 55.0] | 32.6 [24.0 to 42.5] | 37.7 [24.1 to 53.6]
  Female gender | 34.3 [22.5 to 48.5] | 8.2 [4.9 to 13.4] | 13.5 [8.2 to 21.3] | 6.8 [2.7 to 16.1]
  Comorbidities | 10.6 [7.0 to 15.9] | 18.0 [12.5 to 25.4] | 25.0 [17.0 to 35.1] | 17.8 [10.8 to 28.0]
  Baseline laboratory values | 13.2 [8.2 to 20.5] | 15.3 [9.4 to 23.9] | 21.9 [14.4 to 31.9] | 10.5 [4.5 to 22.5]
  Personal experience of chemotherapy regimen risk | 21.4 [13.7 to 31.8] | 16.2 [8.0 to 29.8] | 14.4 [7.1 to 27.0] | 22.6 [12.8 to 36.7]
  Prior chemotherapy | 12.4 [7.6 to 19.5] | 17.0 [11.7 to 24.2] | 14.3 [9.7 to 20.4] | 15.1 [9.4 to 23.4]
  Nutritional status | 4.3 [2.3 to 7.6] | 13.0 [7.8 to 20.8] | 14.3 [7.8 to 24.6] | 11.0 [5.9 to 19.8]
  Planned relative dose intensity | 7.0 [3.4 to 13.9] | 5.7 [2.4 to 13.0] | 10.2 [4.4 to 21.9] | 10.8 [6.0 to 18.8]
  Medications taken | 3.9 [2.2 to 6.9] | 3.2 [1.6 to 6.3] | 11.1 [6.0 to 19.9] | 5.5 [2.2 to 13.1]
  History of prior FN | 4.0 [2.2 to 7.0] | 3.2 [1.6 to 6.3] | 7.0 [3.3 to 14.2] | 2.7 [0.7 to 9.2]
  Documented bone marrow involvement | 1.5 [0.7 to 3.3] | 2.0 [0.8 to 4.8] | 19.4 [11.8 to 30.3] | 1.7 [0.4 to 6.6]
  Prior radiotherapy involving bone marrow | 3.9 [2.3 to 6.6] | 5.9 [3.2 to 10.7] | 2.2 [0.8 to 5.8] | 3.4 [1.2 to 9.2]
  Current infection | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 3.6 [1.8 to 6.9] | 8.8 [4.9 to 15.3] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model.
  Concurrent radiotherapy | 1.2 [0.4 to 3.0] | 2.9 [1.3 to 6.3] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 10.3 [5.4 to 19.0]
  Open wounds | 2.7 [1.3 to 5.4] | 1.4 [0.4 to 4.1] | 3.5 [1.4 to 8.3] | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model.
  Other patient related | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 2.6 [0.9 to 7.1] | 5.0 [2.0 to 11.5] | 2.6 [0.8 to 8.2]
  Other disease/treatment related | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | NA [NA to NA] — Not applicable due to lack of convergence in the statistical model. | 1.1 [0.3 to 4.3] | 2.2 [0.6 to 7.6]

23. Secondary Outcome: Percentage of Participants With an Investigator-assessed FN Risk at or Above the Investigator Self-reported FN-risk Intervention Threshold Who Were Planned to Receive G-CSF PP
Description: At Baseline investigators recorded the FN risk threshold score at which they would use G-CSF PP in their usual clinical practice. For each enrolled participant, the investigator documented their final estimated FN risk score as a percentage based on the participant's medical history and standard of care assessments (their routine practice for assessing this risk), and a decision as to whether G-CSF PP would be administered in Cycle 1.
Time Frame: At Baseline and at enrolment, prior to chemotherapy initiation.
Population: Primary analysis set, participants with investigator-assessed FN risk at or above the investigator FN-risk intervention threshold
Measure: Number; unit: percentage of participants
Arm/Group | At or Above Investigator Threshold
Number analyzed (Participants) | 570
percentage of participants | 82.0

ADVERSE EVENTS:
Description: Adverse Events were not collected for this observational protocol.
Arm/Group | All Enrolled Patients
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.